CLINICAL TRIAL: NCT03137472
Title: Transcranial Magnetic Stimulation (TMS) for Complex Regional Pain Syndrome (CRPS)
Brief Title: TMS for Complex Regional Pain Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Redlich Pain Endowment (Unknown); Rocky Mountain Foundation (Unknown); The Feldman Family Foundation Pain Research Fund (Unknown)
Responsible Party: Principal Investigator, Sean Mackey, Chief, Division of Pain Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25894-3
Record Dates: First submitted 2017-04-28; First posted 2017-05-02 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Complex Regional Pain Syndromes
Keywords: TMS, CRPS, Sham
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single, blinding of participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Treatment (Experimental): Participants will receive active TMS in the target area once daily for two days
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- Sham Treatment (Sham Comparator): Participants will receive active TMS in a non-target area once daily for two days
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — The Magventure TMS stimulator will be used to perform intermittent theta burst followed by high frequency Transcranial Magnetic Stimulation (TMS).

SUMMARY:
The aim of the current study is to assess the efficacy of TMS in the treatment of Complex Regional Pain Syndrome (CRPS). It is hypothesized that participants who receive TMS (Group 1) relative to sham treatment (Group 2) once daily for two days will demonstrate a greater improvement in CRPS-related pain and other associated symptomology (i.e., cognitive, emotional and physical) compared to baseline. Participants will be followed until they reach their baseline for two consecutive weeks to assess safety and duration of symptom alleviation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Diagnosis of CRPS (complex regional pain syndrome) for at least 3 months
* Average pain level reported on Numerical Rating Scale meets entry criteria
* Ability to perform the experimental task and procedures.

Exclusion Criteria:

* MRI contraindication (metal implants or devices, claustrophobia)
* TMS Contraindication (eg metal implant or devices near the site of stimulation)
* History of epilepsy
* History of a psychological or psychiatric disorder that would interfere with study procedures, at the discretion of the researcher.
* Neurologic illness that would interfere with brain integrity
* Current medical condition or medication use that would interfere with study procedures or data integrity, at the discretion of the researcher.
* Currently pregnant or planning to become pregnant.
* On going legal action or disability claim.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-04-24 (Actual); Primary Completion 2026-06-29 (Estimated); Study Completion 2026-06-29 (Estimated)

PRIMARY OUTCOMES:
Change in Pain | 1 week follow-up compared to baseline
  Decrease in CRPS-related Pain Ratings
Duration of Pain Relief | Duration from last treatment until pain returns - up to an estimate of 6 months
  Duration of decreased CRPS-related pain ratings, measured as a length of time until pain returns for two consecutive weeks

SECONDARY OUTCOMES:
Change in Pain-related Symptomology | Duration from last treatment until pain returns - up to an estimate of 6 months
  Decreases in Pain-related Symptomology (i.e., cognitive, emotional and physical)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Pain Management Center, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No